CLINICAL TRIAL: NCT02862444
Title: The Effectiveness of a Culturally Appropriate Intervention for Preventing and Reducing Postpartum Depression Among Arab Women in Southern Israel
Brief Title: A Culturally Appropriate Intervention for Preventing and Reducing Postpartum Depression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Other Study IDs: 0004-16-COM2
Record Dates: First submitted 2016-07-26; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- intervention group: Culturally Appropriate Intervention
  Interventions: Other: Culturally Appropriate Intervention

INTERVENTIONS:
Other: Culturally Appropriate Intervention — Women in the intervention arm will receive a culturally appropriate intervention that will be provided to them according to the five strategies of culturally appropriate interventions of Kreuter et al. (2003).

SUMMARY:
Postpartum depression (PPD) is a highly prevalent and serious mental health problem and is defined as the most recent episode of depression occurring between four weeks and twelve months after childbirth. PPD has negative effects, which are usually strongest during the first six months and may decrease the quality of mother-child interaction, adversely affecting the child's behavior and emotional and cognitive development, as well as the spouse marital relationship.PPD prevalence is estimated at 10 to 20%. A recent studies among Arab-Bedouin women, reported 31% - 43 of PPD.

Aims: To develop and implement a culturally appropriate intervention program by using focus group (FGs) methodology

Methods and Research program description: The study includes two phases. First, qualitative study will be conducted by using focus groups (FGs) method and based on the results of this phase we will develop a culturally based program. The second phase will include implementation and evaluation of the effectiveness of a culturally appropriate intervention.

DETAILED DESCRIPTION:
This study main aim has two aims:

1. To develop and implement a culturally appropriate intervention program by using focus group (FGs) methodology.
2. To evaluate the effectiveness of the culturally appropriate program in preventing PPD among Arab Bedouin women in southern Israel, while taking into consideration different factors.

Methods and Research program description The study includes two phases. First, qualitative study will be conducted by using focus groups (FGs) method and based on the results of this phase the investigators will develop a culturally based program. The second phase will include implementation and evaluation of the effectiveness of a culturally appropriate intervention.

The study first phase Developing a culturally appropriate intervention using focus groups (FGs) At this phase we will conduct four focus groups. Focus Group questions will be designed to encourage participant interaction, and to elicit information relevant to our study aims regarding methods of preventing and reducing PPD among Bedouin women. Three focus groups will take place in the morning as most women do not work. One focus groups will be conducted in the afternoon hours for women who work outside the household.

At the beginning of each FG, the participants will sign an informed consent form, in addition each participant will be asked to complete an anonymous, short demographic questionnaire.

The study second phase Evaluation of the effectiveness of culturally appropriate intervention to prevent PPD. As mentioned above the intervention program will be based on the findings of the FG in the first phase and will take approximately six to nine months and will be conducted in the Arabic language by an Arab research team from the same culture.

Data collection: During the year 2016, women who visit a gynecologist in the women's health center of Clalit in Rahat, Laqqya and Segev-Shalom will be approached by the PhD student and asked to participate in the study.

All women in the intervention and control groups will be screened for PPD symptoms and interviewed face-to-face before the intervention (during pregnancy, beginning at week of 26), four to six weeks postpartum and during three to six months postpartum using a structured questionnaire in Arabic, which will include questions on PPD symptoms, knowledge and attitudes about PPD, and use of mental health care services.

Then group training will be carried out for postpartum women in the intervention arm only.

The interviews will be carried out by the PhD student and other trained female students.

A structured questionnaire in Arabic will be administered, and will include questions on knowledge and attitudes about PPD, PPD symptoms, IPV, self-assessment of health status, chronic diseases and lifestyle behaviors, socio-demographic, socio-economic, and psychological characteristics, obstetrical factors, and use of mental health care services for PPD.

The duration of each interview will be thirty minutes, and the interviews will be conducted in Arabic. Women who report EPDS score of ≥10 will be referred to a family physician, social worker, psychologist and/or a psychiatrist. Question ten on the EPDS refers to thoughts of self-harm, and any positive answer is considered a cause for concern, which means that women who reply positively to question ten, regardless of their EPDS score, will be referred to the nearest mental health service and women that suffer a sever psychiatric condition needing intensive care will be dropped from the study. All women needing help and professional psychiatric counseling will be referred to Dr. Awad-Alktnani, psychiatrist from the same population, which works in Rahat and Soroka Medical Center in Be'er-Sheva, and one of the researchers in the current study.

The study instruments The study instruments will be in Arabic and it will include validated scales and questions that were used in previous research among Arab women in Israel and in Arab countries.

Privacy and Confidentiality of participants and data The first phase of the study: data will be collected anonymously, questionnaires will be saved by the researchers at the university.

In the second phase of the study: participants will sign an informed consent form which include name, social security number, telephone number and a serial number. Informed consent forms will be saved by researchers in Ben-Gurion University in a closed and locked place.

Research tools (questionnaires) will include a serial number only, with no Identifying details of the participants. These questionnaires will also be saved at the university but not in the same folder of the Informed Consent Forms.

For performing statistical analysis: Data will be typed and stored on a computer without identifying details.

Data analysis and statistical methods Statistical analysis of the second phase of the study will be performed using the SPSS statistical software version 20.

Ethical aspects The study (both phases) will start only after approval of the Clalit Health services and Ethics Committee approval

ELIGIBILITY:
Inclusion and exclusion criteria

The study first phase (FGs): will include Arab Bedouin women in southern Israel, aged 18 and over who have experienced childbirth or/and who described themselves as experienced PPD symptoms in the past, could converse in Arabic, are ready to participate in group discussion and could physically attend the group's meetings.

The study second phase (RCT):

Inclusion criteria:

* Arab Bedouin women in southern Israel
* 26-40 weeks of pregnancy
* Without a severe psychiatric or other health condition needing intensive care.

Exclusion criteria:

* Women who do not speak Arabic
* Women who are not of Arab origin
* Women with a severe psychiatric or other health condition needing intensive care

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study includes two phases. First, qualitative study will be conducted by using focus groups (FGs) method and based on the results of this phase the investigators will develop a culturally based program. The second phase will include implementation and evaluation of the effectiveness of a culturally appropriate intervention.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Postpartum depression will be measured by Edinburgh Postnatal Depression Scale (EPDS) | 2016-2018
  Postpartum depression will be measured by Edinburgh Postnatal Depression Scale (EPDS), which was used to identify the high-risk cases of PPD. The EPDS is a ten-item self-rating scale designed to identify PPD and it is widely used in primary care settings. Each item is scored on a three-point scale (from zero to three points), the minimum and maximum total score ranging from 0 to 30, respectively. A score of thirteen and over was found to be the optimal cut-off score for probable major depression. It is accepted to use a score of ten to twelve to indicate low to moderate PPD and a score of ≥13 to indicate probable major PPD.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alfayumi-Zeadna S, Zeadna A, Azbarga Z, Salman L, Froimovici M, Alkatnany A, Grotto I, Daoud N. A Non-Randomized Controlled Trial for Reducing Postpartum Depression in Low-Income Minority Women at Community-Based Women's Health Clinics. Matern Child Health J. 2022 Aug;26(8):1689-1700. doi: 10.1007/s10995-022-03434-1. Epub 2022 Apr 21. PMID 35445883